CLINICAL TRIAL: NCT02904369
Title: Exploratory Pharmacokinetic and Pharmacodynamic Study of Oral F/TAF for the Prevention of HIV Acquisition
Brief Title: PK and PD Study of Oral F/TAF for HIV Prevention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Agility Clinical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A15-137
Record Dates: First submitted 2016-09-01; First posted 2016-09-19 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-01

CONDITIONS: HIV
MeSH Terms: interventions — Emtricitabine; tenofovir alafenamide; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- F/TAF 200/10 (Experimental): Emtricitabine (FTC) + Tenofovir Alafenamide (TAF) (200/10 mg)
  Interventions: Drug: Emtricitabine; Drug: Tenofovir alafenamide
- F/TAF 200/25 (Experimental): Emtricitabine (FTC) + Tenofovir Alafenamide (TAF) (200/25 mg)
  Interventions: Drug: Emtricitabine; Drug: Tenofovir alafenamide
- F/TDF 200/300 (Active Comparator): Emtricitabine (FTC) + Tenofovir Disoproxil Fumarate (TDF) (200/300 mg)
  Interventions: Drug: Emtricitabine; Drug: Tenofovir disoproxil

INTERVENTIONS:
Drug: Emtricitabine
Drug: Tenofovir alafenamide
  Arms: F/TAF 200/10; F/TAF 200/25
Drug: Tenofovir disoproxil
  Arms: F/TDF 200/300

SUMMARY:
This multi-center Phase I study is designed to characterize the PK and PD of F/TAF oral tablets to assess systemic and genital tract bioavailability in healthy women. The oral tablets to be used in the study are F/TAF (200/10 mg), F/TAF (200/25 mg) and F/TDF (200/300 mg, Truvada). Samples will be obtained before, during and after dosing in two study phases.

DETAILED DESCRIPTION:
The purpose of this multi-center Phase I protocol, titled Exploratory Pharmacokinetic and Pharmacodynamic Study of Oral F/TAF for the Prevention of HIV Acquisition is to assess local and systemic pharmacokinetics (PK), pharmacodynamics (PD), and safety characteristics of three oral tablets: F/TAF (200/10 mg), F/TAF (200/25 mg) and F/TDF (200/300 mg).

The study will enroll healthy, non-pregnant, HIV negative, premenopausal women (aged 18-50) who are not at risk of pregnancy and will have two phases: a Single Dose phase (one site only) and a Multiple Dose phase (all three sites).

The enrollment goal is for approximately 72 participants to complete the study. All 72 women are expected to undergo the Multiple Dose phase and the 24 women expected to complete the study at the EVMS site are also expected to undergo the Single Dose phase.

In the Single Dose phase, approximately 24 women will be randomized to one of two products: F/TAF (200/25 mg) or F/TDF (200/300 mg), and will undergo blood, cervicovaginal (CV), and rectal sample collections before and after a single dose for PK and PD assessments. In the Multiple Dose phase, approximately 72 women will be randomized to one of three products: F/TAF (200/10 mg), F/TAF (200/25 mg) or F/TDF (200/300 mg), and will undergo blood, CV, and rectal sample collections for PK and PD assessments before, during and after two weeks of daily dosing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years, inclusive
* General good health (by volunteer history and per investigator judgment) without any clinically significant systemic disease (including, but not limited to significant liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, osteoporosis or bone disease, and diabetes) and with an intact gastrointestinal tract, uterus and cervix.
* History of regular menstrual cycles (for cycling women), by volunteer report
* Estimated calculated creatinine clearance (eCcr) of at least 80 mL/min
* Body Mass Index (BMI) of ≥18 and <35kg/m2; and a total body weight >45 kg (99.2 lbs)
* History of Pap smears and follow-up consistent with standard clinical practice as outlined in the Study Manual or willing to undergo a Pap smear at Visit 1
* Willing to give voluntary consent and sign an informed consent form
* Willing and able to comply with protocol requirements, including swallowing tablets
* May not be using progestin-only hormonal contraception and must be protected from pregnancy by:

  * Condoms
  * Combined hormonal contraceptive (acceptable, but recruitment efforts should be made to limit as much as possible the number of women using them in the study, such that they do not represent the majority of participants.)
  * Copper IUD
  * Sterilization of either partner
  * Heterosexual abstinence
  * Same sex relationship
* If in a relationship, must be in a mutually monogamous relationship with a partner who is not known to be HIV positive and has no known risk of sexually transmitted infections (STIs)

Exclusion Criteria:

* Currently pregnant
* Currently breastfeeding or planning to breastfeed during the course of the study
* History of sensitivity/allergy to any component of the study products, topical anesthetic, or to both silver nitrate and Monsel's solution
* In the last three months, diagnosed with or treated for any STI
* Positive test for Trichomonas vaginalis, Neisseria gonorrhea, Chlamydia trachomatis, HIV, or Hepatitis B surface antigen (HBsAg)
* Symptomatic bacterial vaginosis (BV)
* Current, active Hepatitis C infection
* Chronic or acute vulvar or vaginal symptoms (pain, irritation, spotting/bleeding, discharge, etc.)
* Known bleeding disorder that could lead to prolonged or continuous bleeding with biopsy
* Systemic use in the last two weeks or anticipated use during the study of any of the following: corticosteroids, antibiotics, anticoagulants or other drugs known to prolong bleeding and/or clotting, antifungals, or antivirals or antiretrovirals (e.g. acyclovir, valacyclovir, Viread®, Atripla®, Emtriva®, or Complera®), or drugs that may interact with TAF (e.g., protease inhibitors, anticonvulsants, antimycobacterials, St. John's Wort). See Table 1 from the Patient Information brochure below:
* Current or anticipated chronic use of NSAIDs or Tylenol for the duration of the study
* Positive urine drug screen, or known current drug or alcohol abuse which could impact study compliance. Note: therapeutic use of benzodiazepines is acceptable; investigator may discuss with CONRAD participants that may be eligible for enrollment despite a positive drug screen (e.g., false positives, use of cold medications).
* Participation in any other investigational trial with use of a drug/device within the last 30 days or planned participation in any other investigational with use of a drug/device trial during the study
* Grade 2 or higher laboratory abnormality, per the 2014 update of the Division of AIDS, National Institute of Allergy and Infectious Disease (DAIDS) Table for Grading the Severity of Adverse Events, or clinically significant laboratory abnormality as determined by the clinician
* Abnormal finding on laboratory or physical examination or a social or medical condition in the volunteer which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
Plasma, cervicovaginal and rectal fluid concentrations of tenofovir alafenamide (TAF), tenofovir (TFV), and emtricitabine (FTC) | Day 17
  Concentrations after use of study tablets after single dose, and during (plasma) and after two weeks of daily dosing
PBMC concentrations of tenofovir-diphosphate (TFV-DP), emtricitabine-triphosphate (FTC-TP), deoxyadenosine triphosphate (dATP) and deoxycytidine triphosphate (dCTP) | Day 17
  Concentrations after use of study tablets after single dose, and during and after two weeks of daily dosing
Cervicovaginal tissue concentrations of TAF, TFV, FTC, TFV-DP, FTC-TP, dATP and dCTP | Day 17
  Concentrations after use of study tablets after single dose, and after two weeks of daily dosing
Pharmacokinetic parameter (Cmax) of F/TAF in the systemic compartment | Day 17
  Concentrations after use of study tablets after single dose, and during and after two weeks of daily dosing
p24 antigen production in cervicovaginal and rectal tissue infected with HIV | Day 17
  p24 antigen production in CV tissue infected with HIV ex vivo after a single dose, and in CV and rectal tissue infected with HIV ex vivo after two weeks of daily dosing compared to baseline
Anti-HIV activity in cervicovaginal and rectal fluid (TZM-bl inhibition measured as mean percent reduction compared to control) | Day 17
  Anti-HIV activity in CV and rectal fluid after a single dose, and after two weeks of daily dosing compared to baseline
Pharmacokinetic parameter (Tmax) of F/TAF in the systemic compartment | Day 17
  Concentrations after use of study tablets after single dose, and during and after two weeks of daily dosing
Pharmacokinetic parameter (AUC) of F/TAF in the systemic compartment | Day 17
  Concentrations after use of study tablets after single dose, and during and after two weeks of daily dosing

SECONDARY OUTCOMES:
Number of participants with Grade 2 or higher adverse events | Baseline, Day 17
  Changes from baseline in adverse events

OTHER OUTCOMES:
Anti-HSV activity in cervicovaginal and rectal fluid (mean percentage inhibition of plaque forming units (pfu) in Vero cells infected with HSV-2) | Baseline, Day 17
  Anti-HSV activity in CV and rectal fluid after a single dose, and after two weeks of daily dosing compared to baseline
Number of participants with gastrointestinal adverse events | Baseline, Day 17
  Changes from baseline in adverse events
Number of participants with systemic safety laboratory abnormalities | Baseline, Day 17
  Changes from baseline in safety laboratory abnormalities

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Magee-Womens Research Institute and Foundation, Pittsburgh, Pennsylvania
  - Eastern Virginia Medical School Clinical Research Center, Norfolk, Virginia
- Profamilia, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ouattara LA, Thurman AR, Jacot TA, Cottrell M, Sykes C, Blake K, Fang X, Ju S, Vann NC, Schwartz J, Doncel GF. Genital Mucosal Drug Concentrations and anti-HIV Activity in Tenofovir-Based PrEP Products: Intravaginal Ring vs. Oral Administration. J Acquir Immune Defic Syndr. 2022 Jan 1;89(1):87-97. doi: 10.1097/QAI.0000000000002820. PMID 34878438
- [Derived] Thurman AR, Schwartz JL, Cottrell ML, Brache V, Chen BA, Cochon L, Ju S, McGowan I, Rooney JF, McCallister S, Doncel GF. Safety and Pharmacokinetics of a Tenofovir Alafenamide Fumarate-Emtricitabine based Oral Antiretroviral Regimen for Prevention of HIV Acquisition in Women: A Randomized Controlled Trial. EClinicalMedicine. 2021 May 23;36:100893. doi: 10.1016/j.eclinm.2021.100893. eCollection 2021 Jun. PMID 34041459